CLINICAL TRIAL: NCT06597383
Title: The RApid Switch From 1st Generation Somatostatin Analogues to PaSireOtiDe In Acromegaly ( RAPSODIA )
Brief Title: The RApid Switch From 1st Generation Somatostatin Analogues to PaSireOtiDe In Acromegaly
Acronym: RAPSODIA
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: University of Turin, Italy (Other); University of Padova (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Andrea Giustina, Professor of Endocrinology, IRCCS San Raffaele
Other Study IDs: RAPSODIA
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acromegaly
Keywords: somatostatin analogues; pasireotide; pegvisomant
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, retrospective, national multicenter study aimed to evaluate the impact and efficacy of Time To Switch (TTS) from first-line to second-line medical therapy in Acromegaly.

DETAILED DESCRIPTION:
The study will retrospectively collect clinical, laboratory and anamnestic data of approximately 100 patients evaluated at the UOs involved in the study in last 5 years and 6 months.

Acromegalic patients which neurosurgical intervention was not completely effective or contraindicated or rejected by the patient and for which first-line medical therapy with first-generation somatostatin analogues (octreotide LAR or lanreotide) did not result in disease control and switched to second-line medical therapy will be enrolled. The TTS is the time defined in days and months from the observation that disease is no longer biochemically controlled, defined by the presence of GH levels ≥1 μg/L and IGF-1>1.3×ULN (upper limit of normal), during 1st line therapy, and the start of 2nd line therapy line.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (age ≥ 18 years) affected by acromegaly, including those of childbearing age
* Patients inadequately controlled with first generation somatostatin analogues (GH ≥1 μg/L and IGF-1 >1.3×ULN)
* Second line medical treatment (Pasireotide; Pegvisomant only; combination Pegvisomant + 1st generation SSA) after use of first-line medical treatment
* At least 12 months of follow up during 2nd line therapy
* Signature of the informed consent to the study

Exclusion Criteria:

* age ≤18 years
* Pregnant and/or breastfeeding women
* Patients unable to understand and sign the Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acromegaly treated with second-line medical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of TTS on disease control in acromegalic patients defined by IGF-1 levels <1.3xULN | 12 months
  Retrospective data on biochemical and clinical outcomes of patients affected by acromegaly treated with second-line medical therapy will be collected and analyzed. The patients will be stratified based on the therapeutic switch time (Time To Switch, TTS) < 6 months, between 6 and 12 months and > 12 months, from 1st generation SSA to the different second-line medical approaches (Pasireotide; Pegvisomant alone; Pegvisomant + first generation SSA combination). The impact of TTS on the biochemical and clinical control of illness will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Giustina, Milan, Italy